CLINICAL TRIAL: NCT00212602
Title: ONO-7436 Phase II Study - A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Examine the Efficacy and Safety of ONO-7436 for the Prevention of Cancer Chemotherapy-Induced Nausea and Vomiting in Japan
Brief Title: ONO-7436 Phase II Study in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ONO-7436-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Malignant Tumor
Keywords: ONO-7436, Aprepitant, Vomiting, Nausea
MeSH Terms: conditions — Neoplasms; Vomiting; Nausea | interventions — Aprepitant

INTERVENTIONS:
Drug: ONO-7436

SUMMARY:
The purpose of this study is to examine the efficacy and safety of ONO-7436 for the prevention of cancer chemotherapy-induced nausea and vomiting in patients with malignant tumor

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 20 years or older
2. Patients with malignant tumor who are to be intravenously administered cisplatin as a single dose of 70 mg/m2 or more in under 3 hours
3. Patients whose performance status is 0 to 2
4. Other inclusion criteria as specified in the study protocol

Exclusion Criteria:

1. In case of patients who are previously treated with cisplatin, those having no past history of vomiting as of administration of cisplatin
2. Patients who had vomiting or dry vomiting within 24 hours before the initial administration of the moderate or severe emetic chemotherapy (including cisplatin) on Day 1 of the study
3. Pregnant women, nursing women, women of child-bearing potential, women who wish to become pregnant or women using oral contraception
4. Other exclusion criteria as specified in the study protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2005-08

PRIMARY OUTCOMES:
Patient proportion of complete response (no vomiting and no rescue treatment).

SECONDARY OUTCOMES:
Proportion of patients with no vomiting, no rescue treatment, and no nausea (in each category or combination), frequency of vomiting, and time to first vomiting, and first rescue treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - Chugoku Region Facility, Chugoku
  - Chubu Region Facility, Chūbu
  - Hokkaido Region Facility, Hokkaido
  - Hokuriku Region Facility, Hokuriku
  - Kanto Region Facility, Kanto
  - Kinki Region Facility, Kinki
  - Kyushu Region Facility, Kyushu
  - Shikoku Region Facility, Shikoku
  - Tohoku Region Facility, Tōhoku

REFERENCES:
- [Derived] Takahashi T, Hoshi E, Takagi M, Katsumata N, Kawahara M, Eguchi K. Multicenter, phase II, placebo-controlled, double-blind, randomized study of aprepitant in Japanese patients receiving high-dose cisplatin. Cancer Sci. 2010 Nov;101(11):2455-61. doi: 10.1111/j.1349-7006.2010.01689.x. PMID 20718754